CLINICAL TRIAL: NCT03157310
Title: Bone Metastasis on the Survival of Gefitinib Effective Patients With Non-small Cell Lung Cancer
Brief Title: Bone Metastasis on the Survival of Gefitinib Effective Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-QLH-11
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Overal Survival, Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gefitinib (Experimental): Gefitinib is an selective small molecule epidermal growth factor receptors (EGFRs) tyrosine kinase inhibitors (EGFR-TKI) for non-small cell lung cancer.
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — Daily oral administration of 250 mg Gefitinib
  Other Names: Iressa

SUMMARY:
Gefitinib is a selective small molecule epidermal growth factor receptors (EGFR) tyrosine kinase inhibitors (EGFR-TKI), it's curative effect on non-small cell lung cancer (NSCLC) has been confirmed by a number of prospective clinical trials. The researches aim to analysis whether bone metastasis could affect the survival of NSCLC patients who were effective in Gefitinib treatment over 6 months.

DETAILED DESCRIPTION:
The epidermal growth factor receptors (EGFRs) have inhibitory effects on cell apoptosis, cell growth, angiogenesis and metastasis of tumor cell. The advent of EGFR-TKI significantly improved the clinical efficacy and safety of non-small cell lung cancer (NSCLC) treatment. Compelling study also demonstrate Gefitinib may be effective in the treatment of bone metastases. For NSCLC patients who were effective in EGFR-TKI treatment, whether bone metastasis would shorten the survival time of the patients or reduce the quality of life of patients is worth studying. The researches aim to analysis whether bone metastasis could affect the survival of NSCLC patients who were effective in Gefitinib treatment over 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. histological and (or) cytological diagnosed NSCLC patients.
2. patient was effective in Gefitinib treatment more than 6 months.
3. whether patient received chemotherapy and other treatment is not restricted.
4. whether patient was detected for EGFR gene mutation was not restricted.

Exclusion Criteria:

1. patient with small cell lung cancer.
2. patient without cytology or histopathology diagnosis results.
3. patient with bone metastases cannot rule out other reasons such as inflammation or trauma.
4. patient with poor treatment compliance.
5. patient with incomplete data.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2009-05-01 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2015-07-12 (Actual)

PRIMARY OUTCOMES:
Overal survival of patients | 5 years
  The 5-year survival of NSCLC patients with or without bone metastasis

SECONDARY OUTCOMES:
Survival of patients with both bone metastasis and brain metastasis | 3 years
  Survival of patients with both bone metastasis and brain metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Chun Liu, Dr., Principal Investigator — Qilu Hospital of Shandong University

IPD SHARING:
Plan to Share IPD: No
The patients' data were not allowed to been using outside this research.